CLINICAL TRIAL: NCT05500508
Title: A Phase 1B/2A Study of the Safety, Tolerability and Initial Efficacy of Oral AMXT 1501 Dicaprate and Intravenous Difluoromethylornithine (DFMO) in Patients With Cancer
Brief Title: Oral AMXT 1501 Dicaprate in Combination With IV DFMO
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Required re-formulation of DFMO from IV to capsule to maintain safety
Sponsor: Aminex Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: AMXT1501-102
Record Dates: First submitted 2022-08-10; First posted 2022-08-15 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Cancer; Solid Tumor; Solid Carcinoma; Advanced Cancer; DIPG Brain Tumor; Ovary Cancer; Breast Cancer; Papillary Thyroid Cancer; Head and Neck Cancer; Gastric Cancer; Nsclc; Mesotheliomas Pleural; Mesothelioma Peritoneum; Esophageal Cancer; Diffuse Midline Glioma, H3 K27M-Mutant; Endometrial Cancer; Cervical Cancer; Melanoma; Colorectal Cancer; Glioma, Malignant
Keywords: DFMO IV; AMXT 1501; DFMO
MeSH Terms: conditions — Neoplasms; Diffuse Intrinsic Pontine Glioma; Ovarian Neoplasms; Breast Neoplasms; Thyroid Cancer, Papillary; Head and Neck Neoplasms; Stomach Neoplasms; Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant; Esophageal Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Melanoma; Colorectal Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Escalation (Experimental): Dose escalation of DFMO with AMXT1501 fixed dose will follow a 3 + 3 dose escalation design.
  The AMXT 1501 starting dose administered in the first cohort will be 1200mg total daily dose (200 mg capsules; 3 capsules in morning; 3 capsules in evening) along with IV DFMO administered in continuous infusion at 2mL/hr over a 28 days per cycle. The patient can be treated for additional 28 day treatment cycles as deemed appropriate by their study investigator. Dose escalation of DFMO alone will increase per cohort.
  Interventions: Drug: AMXT1501; Drug: DFMO
- Expansion (Experimental): The expansion cohort will include up to 40 evaluable patients at a proposed RP2D level of AMXT1501 and DFMO defined by AMXT1501-101A study to further characterize safety at proposed RP2D dose level with repeat dosing, and characterize early anti-tumor activity.
  Interventions: Drug: AMXT1501; Drug: DFMO

INTERVENTIONS:
Drug: AMXT1501 — AMXT 1501 dicaprate is D-lys(palmitoyl)-spermine dicaprate salt in 200 mg (free base content) enterically-coated capsules
Drug: DFMO — DFMO is DL-2-(difluoromethyl) ornithine monohydrochloride monohydrate provided as a 200 mg/mL aqueous solution in 20 mL vials.
  Other Names: difluoromethyl ornithine monohydrochloride

SUMMARY:
A Phase 1B/2A study will be conducted to establish safety and dose level of AMXT 1501 dicaprate in combination with IV DFMO, in cancer patients.

DETAILED DESCRIPTION:
The objective of this study is to determine the safety and tolerability of oral AMXT 1501 dicaprate (AMXT1501) in combination with IV DFMO in patients with advanced solid tumors, or DIPG/DMG. Secondary objectives include characterization of plasma pharmacokinetics (PK), pharmacodynamic (PD), and other biomarker efficacy assessments of the impact of AMXT 1501 in combination with IV DFMO on polyamine uptake by circulating lymphocytes (blood cells). To these aims, the study will evaluate the safety, PK, PD, and other biomarker efficacy profiles of orally-administered AMXT 1501 and IV DFMO. Approximately, 56 patients will be enrolled to determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of AMXT 1501 and IV DFMO in combination. The MTD is defined as the highest dose level below at which dose escalation is stopped.

ELIGIBILITY:
INCLUSION CRITERIA

* IMPORTANT NOTE- Younger 12-17 year old patients are also eligible for this study if they meet the noted DIPG or DMG criteria noted below, which is separate from Patient Diagnosed with Advanced Solid Tumors.
* Patients will be eligible for study participation only if they meet ALL the inclusion criteria applicable to their diagnosis.

INCLUSION FOR PATIENTS DIAGNOSED WITH ADVANCED SOLID TUMORS

* Understand and sign written IRB-approved informed consent form and be willing to comply with all study procedures.
* Diagnosed with unresectable, locally advanced, or metastatic solid tumor for which no standard therapy is recognized or for which standard therapy has failed. Planned tumor types for evaluation include:

  * Platinum resistant ovarian cancer (including - primary peritoneal cancer and fallopian tube cancer)
  * Breast cancer
  * Papillary thyroid cancer
  * Head and neck cancer
  * Gastric cancer
  * Non-small cell lung cancer (NSCLC)
  * Mesothelioma: Pleural and peritoneal
  * Esophageal
  * Endometrial cancer
  * Cervical
  * Melanoma
  * Colorectal cancers (colon, rectal)
  * Grade 4 Gliomas (including both IDH WT and IDH-mutant astrocytoma)
* Must be ≥18 years of age.
* Histologically or cytologically documented disease.
* Has evaluable or measurable disease by RECIST v1.1 or mRECIST criteria.

  o For patients with Grade 4 glioma, has evaluable or measurable disease by RANO (Appendix 5).
* Provide tumor tissue from biopsy taken during Screening period.
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) scale.

INCLUSION FOR PATIENTS DIAGNOSED WITH DIPG OR DMG Patients must also meet other generally noted criteria as noted within the protocol

* For patients <18 years of age, the parents or legal guardians must understand and sign the written IRB-approved informed consent form (ICF). The patient, if able, must understand and sign the IRB-approved consent (assent) and be willing to comply with all study procedures.

  o For patients ≥18 years of age, the patient must understand and sign written IRB-approved ICF and be willing to comply with all study procedures.
* Diagnosed with DIPG or DMG.

  o Any anatomic site of origin is acceptable.
* Must be ≥12 years of age and >40 kg in body weight.
* Radiologically documented disease.

  * (a) - Patient with refractory or progressive DIPG or DMG, defined as tumors with a pontine epicenter and diffuse involvement of at least 2/3 of the pons, are eligible without histologic confirmation.
  * (b) - Patients with brainstem tumors that do not meet radiographic criteria or are not considered to be typical DIPG or DMG will be eligible if the tumors have been biopsied and proven to be high-grade gliomas (such as anaplastic astrocytoma, glioblastoma, H3 K27M-mutant DMG).
* Has evaluable or measurable disease by RANO or RAPNO criteria.

  o Has evaluable or measurable disease by RANO (for adults) or RAPNO (for children
* Provide cerebrospinal fluid (CSF) sample. Patients with pontine lesions for whom a radiological diagnosis of DIPG, or DMG is made will be eligible without a CSF sample, although CSF sample is strongly encouraged.
* Performance score:

  * (a) Patients >16 years of age, Karnofsky score ≥50%.
  * (b) Patients ≥12 and ≤16 years of age, Lansky ≥50%. Note: Patients who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

INCLUSION FOR ALL PATIENTS All patients are required to meet these inclusion exclusion criteria to be considered eligible for the study

* Patients must have fully recovered from the acute toxic effects of all prior anti-cancer chemotherapy: The following minimum periods from treatment apply:

  * (a) Myelosuppressive chemotherapy: At least 21 days after the last dose of myelosuppressive chemotherapy (42 days if prior nitrosourea).
  * (b) Hematopoietic growth factors: At least 14 days after the last dose of a long-acting growth factor (e.g., Neulasta) or 7 days for short-acting growth factor.
  * (c) Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur.
  * (d) Immunotherapy: At least 42 days after the completion of any type of vaccination.
  * (e) Monoclonal antibodies: >21 days must have elapsed from the infusion of last dose of antibody and toxicity related to antibody therapy must be recovered to Grade ≤1.
  * (f) Radiation therapy: Patients must have had their last fraction of craniospinal or focal irradiation a minimum of 8-12 weeks prior to enrollment.
  * (g) Stem cell transplant: Patients must be ≥3 months since autologous stem cell transplant. Patients who received allogenic stem cell transplant or solid organ transplant are not eligible for study.
* Patient is able to take oral medications and willing to use an at-home infusion pump.
* Must have adequate bone marrow and renal/hepatic function at the screening and baseline visits, defined as:

  * (a) Absolute neutrophil count (ANC) ≥1.5×109/L without granulocyte colony-stimulating factor (G-CSF) support within 7 days
  * (b) Platelet ≥100×109/L, without transfusion within 7 days
  * (c) Hemoglobin ≥9 g/dL, without transfusion support within 7 days
  * (d) Activated partial thromboplastin time/ partial thromboplastin time (aPTT/PTT) ≤1.5×ULN.
  * (e) Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN (if liver metastases are present, then ≤5×ULN is allowed).
  * (f) Total serum bilirubin ≤1.5×ULN, (except for patients with known Gilbert's Syndrome in whom ≤3×ULN is permitted).
  * (g) The patient is clinically euthyroid.
  * (h) Renal: Serum creatinine <1.5×ULN or creatinine clearance ≥60 mL/min/1.73 m2 for patients with serum creatinine levels >1.5×ULN.
  * (i) Any Grade 3 or higher lab abnormalities should be discussed and approved by the Medical Monitor prior to enrollment (even if not considered clinically significant).
* Active secondary malignancies will not be allowed, with the exception of:

  * (a) Adequately treated basal cell carcinoma, SCC of the skin, or in situ cervical cancer;
  * (b) Adequately treated Stage 1 cancer from which the subject is currently in remission and has been in remission for ≥2 years;
  * (c) Low-risk prostate cancer with Gleason score <7 and prostate-specific antigen <10 ng/mL, or
  * (d) Any other cancer from which the patient has been disease-free for ≥3 years.
* Patient compliance and geographic proximity (as determined by the Principal Investigator [PI]) to allow adequate follow-up.
* Both male and female patients must be willing to consent to using highly effective contraception prior to study entry, while on treatment, and at least 3 months thereafter

EXCLUSION CRITERIA

* Patients will not be eligible for study participation if they meet ANY of the exclusion criteria.
* Please note different criteria for patients with Advanced Solid Tumors (adults) vs patients with DIPG or DMG (pediatric)

EXCLUSION FOR PATIENTS DIAGNOSED WITH ADVANCED SOLID TUMOR(S)

* Have a seizure disorder where >1 seizure has occurred within the last year.
* Patient with treated (surgically excised or irradiated) with stable brain metastases are eligible as long as the treatment was at least 4 weeks prior to initiation of study drug and baseline brain CT with contrast or magnetic resonance imaging (MRI) within 2 weeks of initiation of study drug is negative for new brain metastases. Patients with stable brain metastases must not require therapy with corticosteroids.
* Treatment with radiation therapy, surgery, chemotherapy, or immunotherapy within 4 weeks prior to study entry (6 weeks for nitrosoureas or Mitomycin C). Limited prior palliative radiation may be permissible no less than 2 weeks prior to C1D1 with approval from the Medical Monitor.

EXCLUSION FOR PATIENTS WITH DIPG OR DMG

- Patients with seizure disorders may be enrolled if seizures are well-controlled, defined as no increase in seizure frequency in the prior 7 days.

* Anticonvulsants should be used as clinically indicated.
* The use of enzyme inducing anticonvulsants is not permitted.

EXCLUSION FOR ALL PATIENTS

* Patients with treated (surgically excised or irradiated) stable brain metastases are eligible as long as the treatment was at least 8 to 12 weeks prior to initiation of study drug and baseline brain CT with contrast or MRI within 2 weeks of initiation of study drug is negative for new brain metastases. Patients with brain metastases or who have Grade 4 glioma receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible.
* Have clinically significant cardiovascular disease (e.g., significant cardiac conduction abnormalities, uncontrolled hypertension, myocardial infarction, cardiac arrhythmia or unstable angina, New York Heart Association Grade 3 or greater congestive heart failure, serious cardiac arrhythmia requiring medication, Grade 2 or greater peripheral vascular disease, or history of cerebrovascular accident [CVA]) within 6 months of enrollment.
* History or presence of an abnormal ECG that, in the Investigator's opinion, is clinically meaningful.

  * Screening QTcF interval >480 ms is excluded. In the event that a single QTcF is >480 ms, the patient may enroll if the average QTcF for the 3 ECGs is <480 ms.
  * For patients with an intraventricular conduction delay (QRS interval >120 ms), the JTc interval may be used in place of the QTcF with Sponsor approval. The JTc must be <340 ms if JTc is used in place of the QTcF.
  * Patients with an intraventricular delay due to a left bundle branch block are excluded.

Note: QTcF prolongation due to pacemaker may enroll if the JTc is normal

* Had major surgery, other than diagnostic surgery, within 4-weeks prior to Day 1.
* Have active bacterial, viral, or fungal infections requiring systemic therapy.
* Women who are pregnant or lactating: NOTE: Women of childbearing potential (WOCBP) must have a negative serum pregnancy test within 1 week prior to treatment.

  * Women not OCBP is defined as
  * (i) Postmenopausal with >1 year since last menses

    * -- (a) If <65 years old, follicle-stimulating hormone (FSH) >40 mIU/mL.
    * -- (b) If ≥65 years old and not on hormone replacement therapy (HRT), FSH >30 mIU/mL.
    * -- (c)If ≥65 years old and on HRT, the FSH requirement is not applicable. Postmenopausal females on HRT will be allowed if HRT has been stable for ≥6 months prior to dosing of study drug(s).
  * Written medical documentation of being sterilized (e.g., hysterectomy, double oophorectomy, bilateral salpingectomy) with the procedure performed ≥6 months prior to dosing study drug(s).

Note: Tubal ligation is not considered a form of permanent sterilization.

* Patients may not have any unresolved toxicity >Grade 1 from previous anticancer therapy, except for stable chronic toxicities that are not expected to resolve (i.e., peripheral neuropathy, alopecia, etc.). Patients who have an ongoing requirement for thyroid replacement therapy from prior exposure to a checkpoint inhibitor but who are clinically euthyroid are permitted.
* Have an unwillingness or inability to comply with procedures required in this protocol.
* Current active liver disease from any cause, including hepatitis A (hepatitis A virus immunoglobulin M [Hep A IgM] positive), hepatitis B (hepatitis B virus [HBV] surface antigen positive), or hepatitis C (hepatitis C virus [HCV] antibody positive, confirmed by HCV ribonucleic acid). Patients with HCV with undetectable virus after treatment are eligible. Patients with a prior history of HBV are eligible if quantitative polymerase chain reaction (PCR) for HBV DNA is negative. Note that elevated levels of biotin may interfere with viral serology testing.
* Have a serious nonmalignant disease that, in the opinion of the Investigator or the Medical Monitor, could compromise protocol objectives.
* Patients who are currently receiving any other investigational agent or who have received an investigational agent within the last 28 days, with the exception of any patient who participated in Study AMXT1501-101A.
* Known GI disease or procedure that could interfere with the absorption of study drug, including inability to swallow whole capsules or conditions that may interfere with absorption. The Medical Monitor should be contacted for any questions regarding this exclusion criterion.
* Patients who have exhibited allergic reactions to a similar structural compound, biological agent, or formulation.
* Use of luteinizing hormone-releasing hormone (LHRH) agonist / antagonists are not permitted.
* Use of biotin (i.e., Vitamin B7) or supplements containing biotin higher than the daily adequate intake of 30 µg (NIH-ODS 2020; Section 5.9.2.1). NOTE: Patients who switch from a high dose to a dose of ≤30 µg/day are eligible for study entry.
* Infection with human immunodeficiency virus (HIV)-1 or HIV-2. o Exception: Patients with well-controlled HIV (e.g., CD4 >350/mm3 and undetectable viral load) are eligible.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-12 (Actual)

PRIMARY OUTCOMES:
Determine DLTs and RP2Ds in AMXT 1501 in combination with IV DFMO | 1 year
  Indicate Number of patients with DLTs in AMXT1501 in combination with IV DFMO in patients with advanced cancer to determine the RP2D within the duration of the dose escalation period of the study as defined by the DLT definition of the protocol from baseline to end of Cycle 1
Determine safety and tolerability of AMXT1501 in combination with IV DFMO | 1 year
  To evaluate the safety and tolerability of AMXT1501 and IV DFMO combination in patients through collecting the number of patients with Treatment Related Adverse Events that occur in patients from first dose, AEs assessed by CTCAEv5.0

SECONDARY OUTCOMES:
Determine the PK using AUC of AMXT 1501 and IV DFMO | 6 months
  To evaluate the pharmacokinetics (PK) of AMXT 1501 in combination with IV DFMO in patients
Determine the PK using Cmax of AMXT 1501 and IV DFMO | 6 months
  To evaluate the pharmacokinetics (PK) of AMXT 1501 and IV DFMO
Characterize investigator defined response Overall Response Rate (ORR) using RECIST v1.1 | 6 months
  To characterize Investigator defined Overall Response Rate (ORR) using RECIST v1.1 response criteria.
Characterize investigator defined Duration of Response (DOR) | 6 months
  To characterize Investigator defined Duration of Response (DOR), using RECIST v1.1 response criteria and length of time (in days) from last study drug administration to time patient has progressive disease.
Characterize AMXT1501 and IV DFMO on the expression of immune related gene signatures | 1 year
  Evaluate the effects of AMXT1501 and IV DFMO on the expression of immune related gene signatures, immune cell phenotype by IHC, AMXT1501 and DFMO drug levels impact on polyamine levels

OTHER OUTCOMES:
Evaluate AMXT1501 and DFMO on PD biomarker by evaluating the level/concentration of polyamine uptake. | 6 months
  Will evaluate the effect of AMXT1501 and DFMO on pharmacodynamic (PD) biomarker of polyamine uptake in the blood starting at Cycle 1 through the end of Cycle 2 and again at the beginning of each new cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Sue Lee, MD, Study Chair — Aminex Therapeutics, Inc.; Michael Armstrong, MD, Study Director — IQVIA Biotech
Locations (7):
- United States (6):
  - Mayo Clinic - Arizona, Phoenix, Arizona
  - Mayo Clinic - Florida, Jacksonville, Florida
  - Mayo Clinic - Minnesota, Rochester, Minnesota
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - MD Anderson Cancer Center, Houston, Texas
  - Fred Hutch Cancer Center - Seattle Cancer Care Alliance, Seattle, Washington
- Kids Cancer Centre, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No